CLINICAL TRIAL: NCT05769868
Title: Prospective, Multicenter and Open Study to Evaluate the Efficacy of Esmolol in the Early Identification of Cardiovascular Disorders Induced by Cirrhosis, Diabetes Mellitus and Cardiotoxic Treatments
Brief Title: Efficacy of Esmolol in the Identification of Cardiovascular Disorders by Cirrhosis, Diabetes Mellitus and Cardiotoxic Treatments
Acronym: CIBERbBECHO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: ICI20/00011; 2021-003889-12 (EudraCT Number)
Record Dates: First submitted 2023-02-15; First posted 2023-03-15 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cirrhosis; Diabetes Mellitus; Oncologic Disorders
Keywords: beta blockers; echocardiography; esmolol; systolic function; cardiovascular diagnosis; biomarkers; diagnostic techniques; medical imaging
MeSH Terms: conditions — Fibrosis; Diabetes Mellitus | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): 1 conventional echocardiography without esmolol administration followed by 1 echocardiography with esmolol administration at Baseline and other study visits.
  Interventions: Drug: Esmolol Injection [Brevibloc]

INTERVENTIONS:
Drug: Esmolol Injection [Brevibloc] — Brevibloc® will be administered intravenously by infusion pump following the administration schedule:
  Loading dose of 500 μg/kg for 1 minute, followed by a maintenance infusion of 50 μg/kg/minute over 5 minutes.
  If the target response is not obtained, the loading dose is repeated and the 50 dose is increased by 50 μg/kg/minute to a maximum of 200 μg/kg/minute.
  The objective response to esmolol beta-blockade is defined as a 15-20% reduction in heart rate, with lower limits of 55 bpm and a systolic blood pressure not less than 90 mmHg and diastolic blood pressure not less than 50 mmHg.
  The perfusion is kept active while the echocardiography image acquisition is completed (approx. 15-30 min).
  Other Names: Anatomical Therapeutic Chemical (ATC) code: C07AB09; Esmolol Hydrochloride

SUMMARY:
The purpose of this study is to assess the superiority of esmolol echocardiography over conventional echocardiography in the diagnosis of subclinical myocardial involvement associated with diabetes mellitus 2, cirrhosis and antineoplastic treatments.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 10 days screening period to determine eligibility for study entry. At Baseline, patients who meet the eligibility requirements will be allocate in one of the 4 cohorts according to their medical conditions.

Trial design consists in a Screening period, Baseline, and 6 additional visits until Month-36.

All patients will undergo to a conventional echocardiography and echocardiography with esmolol administration at Baseline. This procedure will be performed at the following visits according their cohort.

Other complementary procedures will be the collection of blood samples to determine biomarkers, as well as hematology and biochemistry, vital signs and another explorations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Absence of previous heart disease, defined as the absence of relevant cardiac structural alterations such as moderate or severe hypertrophy, alteration of segmental contraction, Moderate or severe valvular disease, intraventricular obstructive gradient, or old myocardial infarction.
3. Existence of an at least acceptable ultrasonic window, which allows the visualization of at least 14 of the 17 segments of the LV myocardium.
4. Sinus rhythm, with a basal heart rate greater than 50 bpm.
5. Diabetic patients with a diagnosis of Diabetes Mellitus 2 (DM2) with or without Heart Failure with Normal Ejection Fraction (HFNEF) (n = 300) will be included. Previous diagnosis of HFNEF with clinical stability at the time of inclusion (n = 200). No previous diagnosis of HFNEF (n = 100).
6. 200 patients with cirrhosis stratified by the following additional criteria will be included: Child-Pugh A class (n = 25); Child-Pugh B class (n = 75); Child-Pugh C class (with and without ascites n = 50 and n = 50, respectively).
7. 300 cancer patients will be included, divided into 3 therapeutic groups: 125 patients diagnosed with Lymphoma or Sarcoma receiving chemotherapy based on anthracyclines at high doses (≥ 240 mg / m2); 125 patients with Human Epidermal growth factor Receptor 2 (HER2) positive breast cancer receiving chemotherapy regimen that includes trastuzumab without anthracyclines; 50 patients with hepatocarcinoma receiving treatment with Sorafenib.
8. Expected survival> 6 months, first-diagnosis of cancer, and receiving treatment with chemotherapy that includes any of the previous schemes.
9. A control group (n = 200) without heart disease and without any of the study conditions will be included: diabetes from any cause, cancer or active cancer treatment or some degree of liver disease.

Exclusion Criteria:

1. Contraindication for the administration of esmolol (according to technical data sheet): Hypersensitivity to esmolol hydrochloride; Severe sinus bradycardia (HR <50 bpm); 2nd or 3rd degree atrioventricular block without pacemaker; Cardiogenic shock, severe hypotension, or decompensated heart failure; Untreated pheochromocytoma; Acute asthmatic attack; Concomitant intravenous administration or within the first 48 hours after verapamil.
2. Treatment with beta-blocker drugs (oral, topical or intravenous) in the last 7 days before the study.
3. History of ventricular or supraventricular arrhythmias that prevent the safe withdrawal of antiarrhythmic or braking treatment before the administration of esmolol.
4. History of previous high-grade atrioventricular (AV) conduction disorder in non-pacemaker patients.
5. Severe asthma with bronchial hyperresponsiveness.
6. Patients with acute infection.
7. Participants in other clinical trials in the 30 days prior to the start of the study.
8. Pregnant women, or who plan to be, and women during breastfeeding.
9. Patients with limitation to follow the protocol for any reason.
10. Diagnosis of Diabetes Mellitus (DM) of any type other than type 2 [type 1, Latent Autoimmune Diabetes in Adults (LADA), Maturity-Onset Diabetes of the Young (MODY), New Onset Diabetes After Transplant (NODAT), etc.]
11. Patients in New York Heart Association (NYHA) functional class IV or with advanced heart failure.
12. Treatment with an oral beta-blocker at the time of the examination that cannot be safely temporarily suspended 72 hours before the test.
13. Active evidence of Hepatitis B Virus (HBV) or Hepatitis B Virus (HCV) infection.
14. Personal history of previous cancer requiring systemic treatment (excludes skin or localized cancers treated locally surgically).
15. Previous exposure to systemic antitumor treatment or radiotherapy on the thoracic region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Left Ventricle (LV) ejection fraction | At Baseline (Day 1) until Month-24 according to cohort
  Estimated with 3D echocardiography (Both: convectional and with esmolol administration)
Peak measurement of global LV systolic longitudinal strain | At Baseline (Day 1) until Month-24 according to cohort
  Estimated with 3D echocardiography (Both: convectional and with esmolol administration)
Ejection Intraventricular Pressure Difference (EIVPD) measure | At Baseline (Day 1) until Month-24 according to cohort
  Estimated with M-mode echocardiography (Both: convectional and with esmolol administration)

SECONDARY OUTCOMES:
Ejection fraction | At Baseline (Day 1) until Month-24 according to cohort
  Obtained with 2D echocardiography (Simpson's biplane method)
Interleukin (IL)-1β | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
High-sensitivity IL-6 (hsIL-6) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
Soluble Suppression of Tumorigenicity 2 (ST-2) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
N-terminal fragment of brain natriuretic peptide (NT-proBNP) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
Ultrasensitive troponin I (hsTnI) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
Procollagen type I terminal propeptide (PICP) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
C-terminal telopeptide collagen type I (CITP) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium
Matrix metalloproteinase-1 (MMP-1) | At Baseline (Day 1) until Month-24 according to cohort
  Biochemical variables in blood in relation to the alteration of the different components of the myocardium

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bermejo Thomas, MD, PhD, Principal Investigator — Hospital Universitario Gregorio Marañón
Locations (6):
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia

REFERENCES:
- [Background] Yotti R, Bermejo J, Benito Y, Sanz-Ruiz R, Ripoll C, Martinez-Legazpi P, del Villar CP, Elizaga J, Gonzalez-Mansilla A, Barrio A, Banares R, Fernandez-Aviles F. Validation of noninvasive indices of global systolic function in patients with normal and abnormal loading conditions: a simultaneous echocardiography pressure-volume catheterization study. Circ Cardiovasc Imaging. 2014 Jan;7(1):164-72. doi: 10.1161/CIRCIMAGING.113.000722. Epub 2013 Oct 30. PMID 24173273
- [Background] Yotti R, Bermejo J, Desco MM, Antoranz JC, Rojo-Alvarez JL, Cortina C, Allue C, Rodriguez-Abella H, Moreno M, Garcia-Fernandez MA. Doppler-derived ejection intraventricular pressure gradients provide a reliable assessment of left ventricular systolic chamber function. Circulation. 2005 Sep 20;112(12):1771-9. doi: 10.1161/CIRCULATIONAHA.104.485128. PMID 16172285
- [Background] Yotti R, Ripoll C, Benito Y, Catalina MV, Elizaga J, Rincon D, Fernandez-Aviles F, Bermejo J, Banares R. Left ventricular systolic function is associated with sympathetic nervous activity and markers of inflammation in cirrhosis. Hepatology. 2017 Jun;65(6):2019-2030. doi: 10.1002/hep.29104. Epub 2017 Apr 28. PMID 28195341